CLINICAL TRIAL: NCT01768845
Title: Unrelated Umbilical Cord Blood (UCB) Transplantation
Brief Title: Unrelated Umbilical Cord Blood (UBC)Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU 1909
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Chronic Myelogenous Leukemia (CML); Acute Myelogenous Leukemia (AML); Myelodysplastic Syndrome; Multiple Myeloma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia (CLL); Acute Lymphocytic Leukemia (ALL); Severe Aplastic Anemia
Keywords: Chronic myelogenous leukemia (CML); Acute myelogenous leukemia (AML); Myelodysplastic syndrome; Multiple myeloma; Hodgkin lymphoma; Non Hodgkin lymphoma; Chronic lymphocytic leukemia (CLL); Acute lymphocytic leukemia (ALL); Severe Aplastic Anemia; Cord Blood; Umbilical cord blood transplantation; UBC transplantation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant (Experimental): After a preparative regimen the patient will receive an infusion of one or two umbilical cord blood unit(s) (UBC). The UBC unit(s) will be thawed according to methods of Rubinstein et al. If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for GVHD prophylaxis. On day +30, +60, +100, +180, and +365 the chimeric status of patients will be interpreted by variable number tandem repeat (VNTR) analysis. Immune reconstitution (Digeorge Panel) will also be checked at these time points.
  Interventions: Genetic: umbilical cord blood (UCB)

INTERVENTIONS:
Genetic: umbilical cord blood (UCB) — Infusion will occur after preparative regimen in one or two UCB unit(s). If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for GVHD prophylaxis.

SUMMARY:
Hematopoietic progenitor cell (HPC- primitive cells in the blood, bone marrow and umbilical cord that can restore the bone marrow) transplant can be a curative therapy for the treatment of hematologic malignancies (a disease of the bone marrow and lymph nodes). The source of cells used for the transplant comes from related (sibling) and in cases where there is no sibling match, from unrelated donors through the National Marrow Donor Program. The availability of a suitable donor can be a significant obstacle for patients who need a transplant but do not have a matched donor. Cord blood that has been harvested from an umbilical cord shortly after birth has a rich supply of cells needed for transplant. These stored cord bloods are now being used to transplant adults without a matched donor

Advantages to using cord blood includes a readily available source of cells with no risk to the donor during the collection process, immediate source of cells in urgent situations (no lengthy donor work-up)and a reduction in infectious disease transmission to the recipient.

One of the main disadvantages is the cord blood has a small number of cells needed for transplant. In an adult, usually two cords are needed and large recipients do not qualify because they need too many cells.

This study will use two different preparative regimens (chemotherapy and radiation) followed by one or two umbilical cord units (UBC). The preparative regimen used will be chosen by the physician and is based on patient's age, disease and medical condition at the time of transplant.

Multiple objectives for this study include disease-free and overall survival, treatment related mortality, rate of cells taking hold, and the incidence and severity of the transplant complication called graft versus host disease (GVHD).

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation (allo- HCT) is a curative therapy for the treatment of hematological and non-hematological malignancies and certain non-malignant conditions. Bone marrow or peripheral blood from a Human Leukocyte Antigen (HLA) matched sibling donor is the most commonly used source of allogeneic stem cells. However, HLA matched siblings are available for less than one third of the patients who require allo-Stem Cell Transplant (allo-SCT). In the absence of an HLA matched sibling, volunteer unrelated donors or partially mismatched related donors (PMRD), stored cord blood may be used as a source of allogeneic stem cells. Stored cord blood has been used as a source of allogeneic stem cells in infants and children, but had early skepticism in adults because of concerns about the engraftment potential of the relatively limited number of stem cells. The number of stem cells in a unit of cord blood is generally one log less than the number of stem cells on an average collection of bone marrow from an adult for transplantation.

After the success of the first allogeneic umbilical cord blood transplantation in 1988, programs for banking screened unrelated donor CBSC have been initiated both in the United States and Europe. Dr Pablo Rubenstein started the first such bank at the New York Blood Center (NYBC) in 1993. Since its inception, the NYBC has provided unrelated donor cord blood stem cells for over 1000 transplants. Analysis of outcomes for the initial 562 transplant recipients from the NYBC revealed a cumulative rate of engraftment of 81% by day 42 for PMNs. and 85% by day 180 for platelets. Currently, approximately more than 100,000 cord blood units are available in cord blood banks worldwide and more than 2000 patients have received cord blood transplants from these banks. NetCord, an international cooperative group of cord blood banks, has developed a detailed set of standards for cord blood banking to facilitate international exchanges and to guarantee the quality of these products.

Cord Blood Unit Selection:

UCB units will be required to be a 4 to 6 of 6 HLA-A, -B antigen and -DRB1 allele match with the patient. Typing at HLA-C and -DQ will be obtained but not required in the match strategy. A minimum total nucleated cell (TNC) dose of >2.0 x 107/kg at the time of freezing will be utilized when possible. When using double units, each unit should contain a minimum pre-cryopreserved TNC dose of 1.5 x 107/kg.

UCB Transplant Procedure:

There will be a myeloablative and reduced-intensity preparative regimen that can be given prior to infusion of cord product. The myeloablative approach will be selected in younger patients (<50yo) with a HCT-CI score <3. The reduced-intensity regimen will be selected for all older patients (>50) or younger patients with a hematopoietic cell transplantation-specific comorbidity index (HCT-CI) score >3. The reduced-intensity regimen will also be chosen for any patients being transplanted for indolent/follicular lymphomas, CLL, myeloma, or Hodgkin lymphoma; irrelevant of age or HCT-CI score. On a case by case basis, patients may receive a preparative regimen outside of their designated category as noted above with the approval of the PI, if deemed in the patient's best interest.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-70 years
* Available 4/6, 5/6, or 6/6 HLA antigen match (using A, B, and DRB1) cord blood unit.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Karnofsky greater than or equal to 70%)
* Serum bilirubin less than 2 x upper limit of normal
* Serum creatinine less than 2 mg/dl
* DLCO or FEV1 greater than or equal to 50% predicted
* Left ventricular ejection fraction greater than or equal to 35%
* no uncontrolled infection
* If female, not pregnant
* Informed consent given
* No major organ dysfunction precluding transplantation.
* One of the following malignancies or bone marrow failure syndromes:

  * Chronic myelogenous leukemia (CML)
  * Acute myelogenous leukemia (AML)
  * Myelodysplastic syndrome
  * Multiple myeloma
  * Hodgkin lymphoma
  * Non-Hodgkin lymphoma
  * Chronic lymphocytic leukemia (CLL)
  * Acute lymphocytic leukemia (ALL)
  * Severe Aplastic Anemia

Exclusion Criteria:

* Patient pregnant
* Age less than 16, greater than 70
* ECOG performance status of greater than 2 (Karnofsky less than 70%)
* Psychiatric disorder or mental deficiency of the patient sufficiently severe as to make compliance with the BMT treatment unlikely, or making informed consent impossible
* Serum bilirubin greater than or equal to 2 x upper limit of normal, transaminases greater than 3 x upper limit of normal
* Serum creatinine greater than or equal to 2 mg/dl
* DLCO less than 50% predicted
* Left ventricular ejection fraction less than 35%
* Major anticipated illness or organ failure incompatible with survival from Bone Marrow Transplant (BMT)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Craig, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospitals Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant: After a preparative regimen the patient will receive an infusion of one or two umbilical cord blood unit(s) (UBC). The UBC unit(s) will be thawed according to methods of Rubinstein et al. If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for graft versus host disease (GVHD) prophylaxis. On day +30, +60, +100, +180, and +365 the chimeric status of patients will be interpreted by VNTR analysis. Immune reconstitution (Digeorge Panel) will also be checked at these time points.
  umbilical cord blood (UCB): Infusion will occur after preparative regimen in one or two UCB unit(s). If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for GVHD prophylaxis.
Period: Overall Study
Arm/Group | Transplant
Started | 34
Completed | 11
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Transplant
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: Defined as neutrophil recovery associated with donor engraftment within the first 60 days of transplant
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Transplant: After a preparative regimen the patient will receive an infusion of one or two umbilical cord blood unit(s) (UBC). The UBC unit(s) will be thawed according to methods of Rubinstein et al. If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for GVHD prophylaxis. On day +30, +60, +100, +180, and +365 the chimeric status of patients will be interpreted by VNTR analysis. Immune reconstitution (Digeorge Panel) will also be checked at these time points.
  umbilical cord blood (UCB): Infusion will occur after preparative regimen in one or two UCB unit(s). If two products are used, they will be administered sequentially on the same day 1-6 hours apart. Tacrolimus and mycophenolate mofetil (MMF) will be used for GVHD prophylaxis.
Arm/Group | Transplant
Number analyzed (Participants) | 34
Participants | 29

2. Secondary Outcome: Overall Survival at Day 180 Post-transplant
Description: Number of Participants with Overall survival at day 180 transplant.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant
Number analyzed (Participants) | 34
Participants | 18

ADVERSE EVENTS:
Time Frame: 6 months
Description: Systematic assessment of adverse events was completed through that participants all being followed per routine schedule for transplant patients with regular examinations by their care provider with adverse event discovery per standard assessment.
Arm/Group | Transplant
All-Cause Mortality (participants affected / at risk) | 21/34
Serious Adverse Events (participants affected / at risk) | 1/34
Other Adverse Events (participants affected / at risk) | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant (N=34)
Infection (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT01768845/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT01768845/ICF_001.pdf